CLINICAL TRIAL: NCT04823260
Title: A Multi Center Two Part Study to Evaluate the Efficacy and Safety of NMN as an Anti-ageing Supplement in Middle Aged and Older (40-65 Years) Adults
Brief Title: To Evaluate the Efficacy and Safety of NMN as an Anti-ageing Supplement in Middle Aged and Older (40-65 Years) Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abinopharm, Inc (Network)
Collaborators: ProRelix Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: AP-NMN-CT01-21
Record Dates: First submitted 2021-03-06; First posted 2021-03-30 (Actual); Last update posted 2021-10-01 (Actual); Status verified 2021-09

CONDITIONS: Aging
Keywords: Nicotinamide Mononucleotide (NMN); Anti Ageing; Telomerase
MeSH Terms: interventions — Nicotinamide Mononucleotide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Arm A = 300 mg NMN supplement (n = 20) (Active Comparator): Subjects who are assigned to 300 mg arm (NMN) will be instructed to take 2 capsules after breakfast once a day with ambient temperature water for 60 days.
  Interventions: Drug: Nicotinamide Mononucleotide
- Arm B = Placebo 300 mg (n=07) (Placebo Comparator): Subjects who are assigned to 300 mg arm (placebo) will be instructed to take 2 capsules after breakfast once a day with ambient temperature water for 60 days.
  Interventions: Other: Placebo
- Arm C = NMN Supplement 600 mg (n= 20) (Active Comparator): Subjects who are assigned to 600 mg arm (NMN) will be instructed to take 4 capsules after breakfast once a day with ambient temperature water for 60 days.
  Interventions: Drug: Nicotinamide Mononucleotide
- Arm D = Placebo 600 mg (n=07) (Placebo Comparator): Subjects who are assigned to 600 mg arm (Placebo) will be instructed to take 4 capsules after breakfast once a day with ambient temperature water for 60 days.
  Interventions: Other: Placebo
- Arm E = NMN Supplement 900 mg (n=10) (Active Comparator): Subjects who are assigned to 900 mg arm (NMN) will be instructed to take 6 capsules after breakfast once a day with ambient temperature water for 60 days.
  Interventions: Drug: Nicotinamide Mononucleotide
- Arm F = Placebo 900 mg (n=06) (Placebo Comparator): Subjects who are assigned to 900 mg arm (Placebo) will be instructed to take 6 capsules after breakfast once a day with ambient temperature water for 60 days.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Nicotinamide Mononucleotide — Nicotinamide adenine dinucleotide (NAD+) is an essential cofactor in all living cells involved in fundamental biological processes. Depletion in the levels of NAD+ is associated with traits of aging, many age-related diseases like cancer, metabolic disorders and neurological disorders. Evidence stemming from recent studies have unveiled numerous roles of NAD+ metabolism on aging and longevity and delaying the progression of age-related diseases
  Arms: Arm A = 300 mg NMN supplement (n = 20); Arm C = NMN Supplement 600 mg (n= 20); Arm E = NMN Supplement 900 mg (n=10)
Other: Placebo — Rice flour in white capsule resembling NMN
  Arms: Arm B = Placebo 300 mg (n=07); Arm D = Placebo 600 mg (n=07); Arm F = Placebo 900 mg (n=06)

SUMMARY:
It will be a two-part study. Part I will be six arms; randomized, double blind, parallel design, placebo-controlled dose ranging study. Part II will be open-label single dose study at the highest dose.

A total of 90 Subjects (Part 1 & Part 2) will be enrolled in the study. The Part 1 group subjects (80 Subjects) shall be randomly distributed between the six arms, i.e. 20 Subjects each in IP arms, and 7, 7 and 6 subjects in corresponding placebo arms.

All Part 2 Group subjects (10 Subjects) will be assigned into the cluster where all receive the maximum NMN dose (900 mg)

DETAILED DESCRIPTION:
It will be a two-part study. Part I will be six arms; randomized, double blind, parallel design, placebo-controlled dose ranging study. Part II will be open-label single dose study at the highest dose.

Total number of Subjects is N = 90 (Part 1 & Part 2) Part I: six arms Arm A = 300 mg NMN supplement (n = 20) Arm B = Placebo of 300 mg NMN supplement (n = 07) Arm C = 600 mg NMN supplement (n = 20) Arm D = Placebo of 600 mg NMN supplement (n = 07) Arm E = 900 mg NMN supplement (n = 20) Arm F = Placebo of 900 mg NMN supplement (n = 06) Part II 900 mg NMN supplement (n = 10) Duration of Protocol Therapy = 60 Days Study Population= Middle aged or older male or female subjects (40-65 years)

The duration of each subject's participation in the study will be of 60 days. Scheduled study visits will include:

* Visit 1 (Screening, Day -4)
* Visit 2 (Baseline/Randomization visit, Day 1)
* Visit 3 (Day 30).
* Visit 4 (End of study, Day 60) A window (± 2 days) will be considered acceptable for each scheduled visit following the baseline visit.

During Visit 1 (Screening), informed consent will be obtained before any study procedures take place. After subject has consented, medical history will then be documented, including the concomitant medications (if any). Physical examination and ECG will be carried out for all subjects. Subjects' vital signs will be recorded along with pulse pressure (PP). Their laboratory investigations like Hematology, Clinical chemistry and Urinalysis will be done. They will be symptomatically assessed for COVID-19. They shall undergo the screening procedure by inclusion and exclusion criteria. Subject's demography data will be collected. They will be given instructions for the next visit.

At Visit 2 (Day 1, Baseline visit), eligibility confirmation will be done, and each enrolled subject will be randomly assigned in double-blind fashion, in 1:1 ratio to the test product or the Placebo or to the maximum dose group (Part 2 subjects). Blinded investigational product will be dispensed to subjects for Part 1 who meet all the inclusion and none of the exclusion criteria. Part 2 group subjects will be dispensed with maximum dose of NMN (900mg) without any blinding. Subjects will be instructed to take two to six capsules (depending on thegroups that the subjects fall under) of the either placebo or NMN once a day with ambient temperature water before breakfast. They shall be recording the dosing details in subject diaries. The Investigational Product will be taken by the subject at home right from the first dose. Subjects will be evaluated through SF-36 questionnaire for their health. They will be required to answer the list of questions pertaining to their health. (PI, CRC or site staff will fill SF-36 questionnaire in visit 2, 3 and 4 by asking the subject). All the baseline assessments for efficacy will be performed.

At visit 3 (Day 30) and visit 4 (Day 60), subjects will return to the clinic to review and collect subjects' diaries, safety data and medication reconciliation. Efficacy and safety assessments will be done at both the visits.

Subjects will be asked to bring their subject diaries and used/unused Investigational Product every time they visit the site(empty bottles in case of used IP). Enough quantity of Investigational Product will be dispensed every visit. Subjects' vital signs will be recorded along with pulse pressure (PP) at all visits. Adverse event assessment and concomitant assessment will be done at each visit along with compliance with study supplement administration.

End points:

Primary efficacy endpoints (Part I ) Blood cellular NAD/NADH concentration in serum [ Time Frame: Baseline, 1 month and 2 Months] Six minutes walking endurance test [ Time Frame: Baseline, 1 month and 2 Months] SF-36 questionnaire [ Time Frame: Baseline, 1 month and 2 Months]

Secondary endpoints :

1. To compare the safety of NMN versus placebo [ Time Frame: Baseline to 2 Months]
2. Monitoring and documentation of number and type of adverse events including changes on laboratory parameter (blood chemistry, lipid profile, LFT and RFT)
3. To compare the tolerability of NMN versus placebo [ Time Frame: Baseline to 2 Months] Tolerability: Number of participants that dropout due to adverse events including lab values
4. Monitoring and documentation of subject dropout due to adverse events
5. To compare the safety of the different NMN doses [ Time Frame: Baseline to 2 Months]
6. Monitoring and documentation of number and type of adverse events including changes on laboratory parameter (blood chemistry, lipid profile, LFT and RFT)
7. To compare the tolerability different NMN doses [ Time Frame: Baseline to 2 Months] Tolerability: Number of participants that dropout due to adverse events including lab values Monitoring and documentation of subject

Exploratory endpoints :

1. BMI
2. HOMA (Homeostatic model assessment) Biological Age using Aging.Ai 3.0 calculator [ Time Frame: Baseline to 2 Months]

Primary Endpoints : (Part II)

Evaluation will include the following parameters:

1. Telomerase test results [ Time Frame: Baseline and 2 Months]
2. SF-36 questionnaire [ Time Frame: Baseline and 2 Months]

Secondary endpoint:

1. Safety of NMN [ Time Frame: Baseline to 2 Months]
2. Monitoring and documentation of number and type of adverse events including changes on laboratory parameter (blood chemistry, lipid profile, LFT and RFT, CEA test)

ELIGIBILITY:
Inclusion Criteria: (Applicable to both parts)

1. Male/females of 40 to 65 years of age
2. Body Mass Index (BMI) between 18.5 and 35 kg/m2
3. Able to provide written Informed Consent
4. Able to follow verbal and written study directions
5. Must not be taking or be willing to take any supplements containing any form of niacin for seven days prior to baseline and for the duration of the study.
6. Able to maintain consistent diet and lifestyle habits throughout the study
7. Male and female subjects must be willing to agree to use effective contraceptive methods while on treatment and for 3 months after the completion of study
8. Willing to consume assigned supplement (NMN or placebo) for 2 months

Exclusion Criteria: (Applicable to both parts).

1. Participants on current use of prescription or over-the-counter nicotinic acid
2. Use of statin drugs
3. Having used any tobacco product or used a recreational drug in the past 6 months
4. Having abnormal screening laboratory test values or other lab test result(s) that would preclude study participation in the judgment of the investigator
5. Documented presence of atherosclerotic disease and/or cardiopulmonary disease
6. History of drug or alcohol abuse
7. History of unstable depression or mental illness within the last 6 months for which the investigator believes could impact the participant's ability to comply with study requirements
8. Unwilling to discontinue use of conventional multivitamin/mineral or other supplements at least two weeks prior to the study start
9. Participating in or planning to begin a weight loss diet during the study period,
10. Lifestyle or schedule incompatible with the study protocol
11. Known hypersensitivity to any form of niacin used during the study
12. Women with positive result for Urine Pregnancy Test or gestation period or breastfeeding
13. Other diseases or medications, according to the investigator, that would interfere directly in the results of the study or jeopardize the health of the participant.
14. Currently, or within the past 30 days, enrolled in a different clinical investigation
15. Inability to provide a venous blood sample
16. Unable or unwilling to provide written informed consent for participation in study

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2021-05-25 (Actual); Primary Completion 2021-09-09 (Actual); Study Completion 2021-09-09 (Actual)

PRIMARY OUTCOMES:
Blood cellular NAD+/ NADH | Baseline
  Blood cellular NAD+ / NADH concentration in serum
Blood cellular NAD+/ NADH | 1 month
  Blood cellular NAD+ / NADH concentration in serum
Blood cellular NAD+/ NADH | 2 month
  Blood cellular NAD+ / NADH concentration in serum
Six walking endurance test | Baseline
  Six minutes walking endurance test
Six walking endurance test | 1 month
  Six minutes walking endurance test
Six walking endurance test | 2 month
  Six minutes walking endurance test
SF-36 questionnaire | Baseline
  Short Form-36 questionnaire is a general health questionnaire consisting of 36 questions. The quality of life among the study participants using questionnaire by comparing with end of study.
SF-36 questionnaire | 1 month
  Short Form-36 questionnaire is a general health questionnaire consisting of 36 questions. The quality of life among the study participants using questionnaire by comparing with end of study.
SF-36 questionnaire | 2 month
  Short Form-36 questionnaire is a general health questionnaire consisting of 36 questions. The quality of life among the study participants using questionnaire by comparing with end of study.
PART II : Telomerase test results | Baseline
  Telomere are repetitive nucleotide elements at the end of chromosomes that protect chromosomes from degradation and genetic information loss.In this study we will be doing absolute Human telomere length quantification qPCR assay using a RUO commercial kit. The method uses delta Cq method for calculating relative telomere length with reference DNA used.
PART II : Telomerase test results | 2 Months
  Telomere are repetitive nucleotide elements at the end of chromosomes that protect chromosomes from degradation and genetic information loss.In this study we will be doing absolute Human telomere length quantification qPCR assay using a RUO commercial kit. The method uses delta Cq method for calculating relative telomere length with reference DNA used.
PART II : SF-36 questionnaire | Baseline
  Short Form-36 questionnaire is a general health questionnaire consisting of 36 questions. The quality of life among the study participants using questionnaire by comparing with end of study.
PART II : SF-36 questionnaire | 2 months
  Short Form-36 questionnaire is a general health questionnaire consisting of 36 questions. The quality of life among the study participants using questionnaire by comparing with end of study.

SECONDARY OUTCOMES:
safety of NMN | Baseline
  To compare the safety of NMN versus placebo
safety of NMN | 2 Months
  Monitoring and documentation of number and types of adverse events including changes on laboratory parameter (blood chemistry, lipid profile, LFT and RFT)
Tolerability of NMN | Baseline
  Number of participants that drop out due to adverse events including lab values. Monitoring ad documentation of subject drop out due to adverse events.
Tolerability of NMN | 2 months
  Number of participants that drop out due to adverse events including lab values. Monitoring ad documentation of subject drop out due to adverse events.
Safety of the different NMN doses | 2 Months
  Monitoring and documentation of number and types of adverse events including changes in lab parameter (blood chemistry, lipid profile, LFT, RFT)
Tolerability different NMN doses | Baseline
  Number of participants that drop out due to adverse events including lab values
Tolerability different NMN doses | 2 Months
  Number of participants that drop out due to adverse events including lab values
PART II : Safety of NMN | Baseline
  Monitoring and documentation of number and types of adverse events including changes in lab parameter (blood chemistry, lipid profile, LFT, RFT)
PART II : Safety of NMN | 2 Months
  Monitoring and documentation of number and types of adverse events including changes in lab parameter (blood chemistry, lipid profile, LFT, RFT)

OTHER OUTCOMES:
BMI | Baseline
  Body Mass Index (BMI) is a person's weight in kilograms divided by the square of height in meters. A high BMI can be an indicator of high body fatness.
BMI | 2 months
  Body Mass Index (BMI) is a person's weight in kilograms divided by the square of height in meters. A high BMI can be an indicator of high body fatness.
HOMA (Homeostatic model assessment) | Baseline
  Homeostatic model assessment (HOMA) is a method for assessing β-cell function and insulin resistance (IR) from basal (fasting) glucose and insulin or C-peptide concentrations.
HOMA (Homeostatic model assessment) | 2 months
  Homeostatic model assessment (HOMA) is a method for assessing β-cell function and insulin resistance (IR) from basal (fasting) glucose and insulin or C-peptide concentrations.
Biological Age using Aging.Ai 3.0 calculator | Baseline
  Biological age, also referred to as physiological age, takes many lifestyle factors into consideration, including diet, exercise and sleeping habits, to name a few.
Biological Age using Aging.Ai 3.0 calculator | 2 Months
  Biological age, also referred to as physiological age, takes many lifestyle factors into consideration, including diet, exercise and sleeping habits, to name a few.

CONTACTS AND LOCATIONS:
Overall Officials: Mr.Lin Yi, Study Chair — Abinopharm, Inc
Locations (2):
- India (2):
  - Swasthiya Clinic and Research Center, Pune, Maharashtra
  - Sunad Ayurved, Pune, Maharashtra

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yi L, Maier AB, Tao R, Lin Z, Vaidya A, Pendse S, Thasma S, Andhalkar N, Avhad G, Kumbhar V. The efficacy and safety of beta-nicotinamide mononucleotide (NMN) supplementation in healthy middle-aged adults: a randomized, multicenter, double-blind, placebo-controlled, parallel-group, dose-dependent clinical trial. Geroscience. 2023 Feb;45(1):29-43. doi: 10.1007/s11357-022-00705-1. Epub 2022 Dec 8. PMID 36482258